CLINICAL TRIAL: NCT01805037
Title: A Phase I-II Trial of Brentuximab Vedotin Plus Rituximab as Frontline Therapy for Patients With CD30+ and/or EBV+ Lymphomas
Brief Title: Brentuximab Vedotin + Rituximab as Frontline Therapy for Pts w/ CD30+ and/or EBV+ Lymphomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Northwestern University (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Principal Investigator, Barbara Pro, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 12H09; NCI-2012-03090 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00072695 (Other: Northwestern University IRB#)
Record Dates: First submitted 2013-02-27; First posted 2013-03-05 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Epstein-Barr Virus Infection; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Progressive Hairy Cell Leukemia, Initial Treatment; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage IA Mycosis Fungoides/Sezary Syndrome; Stage IB Mycosis Fungoides/Sezary Syndrome; Stage II Adult Hodgkin Lymphoma; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IIA Mycosis Fungoides/Sezary Syndrome; Stage IIB Mycosis Fungoides/Sezary Syndrome; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IIIA Mycosis Fungoides/Sezary Syndrome; Stage IIIB Mycosis Fungoides/Sezary Syndrome; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Stage IVA Mycosis Fungoides/Sezary Syndrome; Stage IVB Mycosis Fungoides/Sezary Syndrome; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Untreated Hairy Cell Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Epstein-Barr Virus Infections; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, Large B-Cell, Diffuse; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Brentuximab Vedotin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (brentuximab vedotin, rituximab) (Experimental): INDUCTION: Patients receive brentuximab vedotin IV over 30 minutes once weekly for 3 weeks and rituximab IV once weekly for 4 weeks. Patients unable to achieve CR may receive additional optional consolidation therapy identical to induction therapy.
  MAINTENANCE THERAPY: Patients receive brentuximab vedotin IV once every 3 weeks and rituximab IV once every 6 weeks. Treatment repeats every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: brentuximab vedotin; Biological: rituximab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: brentuximab vedotin — Given IV
  Other Names: Adcetris; anti-CD30 ADC SGN-35; anti-CD30 antibody-drug conjugate SGN-35; antibody-drug conjugate SGN-35; SGN-35
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of this study is to evaluate how safe and effective the combination of two different drugs (brentuximab vedotin and rituximab) is in patients with certain types of lymphoma. This study is for patients who have a type of lymphoma that expresses a tumor marker called CD30 and/or a type that is associated with the Epstein-Barr virus (EBV-related lymphoma) and who have not yet received any treatment for their cancer, except for dose-reduction or discontinuation (stoppage) of medications used to prevent rejection of transplanted organs (for those patients who have undergone transplantation). This study is investigating the combination of brentuximab vedotin and rituximab as a first treatment for lymphoma patients

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of brentuximab vedotin and rituximab in patients with lymphoid malignancies that are cluster of differentiation (CD) 30 positive (+) and/or Epstein-Barr virus (EBV)+, and to determine the recommended phase 2 dose (RP2D) of the combination. (Phase I) II. To evaluate the efficacy, as measured by response rates, of brentuximab vedotin and rituximab in patients with lymphoid malignancies that are CD30+ and/or EBV+. (Phase II)

SECONDARY OBJECTIVES:

I. To further evaluate the frequency and severity of toxicity. (Phase II) II. To further evaluate the clinical efficacy of the combination of brentuximab vedotin and rituximab, as measured by progression free survival (PFS) and overall survival (OS) at one year after the end of treatment. (Phase II) III. To determine the effects of the combination of brentuximab vedotin and rituximab on markers of EBV activation and proliferation. (Phase II) IV. Further evaluate efficacy as measured by time to cytotoxic chemotherapy. (Phase II) V. Further evaluate efficacy as measured by observed rates of graft rejection. (Phase II)

TERTIARY OBJECTIVES:

I. To determine whether and to what extent CD30 expression predicts for response and outcome.

II. To determine whether and to what extent expression of EBV markers predicts for response and outcome.

III. To determine whether changes in serum levels of EBV correlate with response and subsequent loss of response to therapy.

OUTLINE: This is a phase I, dose-escalation study of brentuximab vedotin followed by a phase II study.

INDUCTION: Patients receive brentuximab vedotin intravenously (IV) over 30 minutes once weekly for 3 weeks and rituximab IV once weekly for 4 weeks. Patients unable to achieve complete remission (CR) may receive additional optional consolidation therapy identical to induction therapy.

MAINTENANCE THERAPY: Patients receive brentuximab vedotin IV once every 3 weeks and rituximab IV once every 6 weeks. Treatment repeats every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD30+ and/or EBV+ lymphoid malignancy; in addition, there must be evidence of CD20 expression (at any level)
* In cases of post-transplant lymphoproliferative disorder (PTLD) arising in patients who are pharmacologically immunosuppressed, reduction of immunosuppression (RI) must be attempted prior to or in conjunction with enrollment, with the exception of those for whom RI would pose excessive threat of clinically significant graft rejection (as judged by local investigator)
* No prior chemotherapy or radiotherapy for PTLD or diffuse large B-cell lymphoma (DLBCL), with the exception of corticosteroids for 10 or fewer days at any dose (no washout period required)
* No prior surgical intervention, unless performed for the sake of tissue diagnosis or on an urgent basis for disease-related threat to life, limb, or organ function
* Bi-dimensionally measurable disease (at least 1 cm)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 750/mcL
* Platelets >= 50,000/mcl
* Total bilirubin =< 2 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum pyruvate glutamate transaminase [SPGT]) =< 3 X institutional ULN
* Creatinine =< 2 X institutional ULN
* NOTE: Patients who do not meet the above criteria because of disease involvement of the organ in question, or because of acute systemic illness due to lymphoma, may enroll with permission of the study Principal Investigator (PI) and approval from the Data Monitoring Committee; this flexibility be allowed due to the heterogeneity of the patient population, the wide range of complications seen in the initial presentation of EBV-related malignancy, and the frequent difficulty encountered in attempting to clearly document that organ dysfunction is the result of an underlying lymphoproliferative disorder
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Patients must be free of any prior malignancies for >= 1 year; NOTE: the exception to this would be currently treated squamous cell and basal cell carcinoma of the skin, carcinoma in situ of the cervix, breast, or bladder, or surgically removed melanoma in situ of the skin (stage 0) with histologically confirmed free margins of excision; in addition, it is well-recognized that patients at highest risk for EBV-related lymphoma (ie, those with chronic immunosuppression) are also at high risk for various malignancies, both invasive and non-invasive; therefore, exceptions may also be granted on a case-by-case basis, at the discretion of the PI with approval from the Data Monitoring Committee, for those patients with good clinical control of active malignancy, if the EBV-related lymphoma is considered to be a more immediate threat to the subject's health and/or life
* Ability to understand and the willingness to sign a written informed consent; all patients must have signed, witnessed informed consent prior to registration

Exclusion Criteria:

* Chemotherapy (including monoclonal antibodies) or radiotherapy, administered for any condition, within 4 weeks prior to entering the study or incomplete recovery from adverse events due to agents administered more than 4 weeks earlier
* Ongoing treatment with any other investigational agents
* Known central nervous system (CNS) involvement of lymphoma
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to brentuximab vedotin and/or rituximab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known human immunodeficiency virus (HIV) infection
* Known John Cunningham (JC) virus infection and/or progressive multifocal leukoencephalopathy (PML)
* Clinically active hepatitis A, B, or C infections; NOTE: patients with chronic hepatitis C (HCV) or hepatitis B (HBV) infection may enroll if other laboratory criteria are met; those with HBV surface antigen positivity may enroll only if maintained on appropriate suppressive antiviral therapy, per treating investigator's discretion, for the duration of enrollment in the trial
* Pregnancy or active nursing of an infant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Petrich, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tufts University School of Medicine, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on March 4th, 2013 with goal of up to 33 patients. The 1st patient started treatment in Phase 1 on March 5th, 2013. 6 patients were accrued in Phase 1. March 26th, 2014 the study opened to Phase II, 14 patients were accrued. October 29th, 2018 the study closed due to lack of funding.
Groups:
- Brentuximab Vedotin Dose Level -1 (0.8 mg/kg): Treatment:
  Induction:
  * Brentuximab vedotin 0.8 mg/kg IV infusion over 30 minutes, weekly x 3 (1 cycle = 4 weeks )
  * Rituximab 375 mg/m2 IV infusion per standard protocol, once weekly for 4 weeks (1 cycle = 4 weeks)
  Consolidation (optional): Identical to Induction.
  Maintenance: Brentuximab vedotin 1.8 mg/kg IV infusion over 30 minutes once every 3 weeks (1 cycle = 3 weeks), for a total of one year from the first induction dose or until progression of disease. Rituximab 375 mg/m2 IV infusion per standard protocol, once every 6 weeks for a total of one year from the first induction dose or until progression of disease.
- Brentuximb Vedotin Dose Level 1 (1.2 mg/kg): Induction:
  * Brentuximab vedotin 1.2 mg/kg IV infusion over 30 minutes, weekly x 3 (1 cycle = 4 weeks
  * Rituximab 375 mg/m2 IV infusion per standard protocol, once weekly for 4 weeks (1 cycle = 4 weeks)
  Consolidation (optional): Identical to Induction.
  Maintenance:
  * Brentuximab vedotin 1.8 mg/kg IV infusion over 30 minutes once every 3 weeks (1 cycle = 3 weeks), for a total of one year from the first induction dose or until progression of disease.
  * Rituximab 375 mg/m2 IV infusion per standard protocol, once every 6 weeks for a total of one year from the first induction dose or until progression of disease.
Period: Induction (4 Weeks)
Arm/Group | Brentuximab Vedotin Dose Level -1 (0.8 mg/kg) | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Started | 0 | 20
Received Dose of Study Drug | 0 | 20
Completed | 0 | 20
Not Completed | 0 | 0
Period: Consolidation (Optional, 4 Weeks)
Arm/Group | Brentuximab Vedotin Dose Level -1 (0.8 mg/kg) | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Started | 0 | 6 (Consolidation is optional for patients who have a partial or complete response during induction.)
Received Dose of Study Drug | 0 | 6
Completed | 0 | 6
Not Completed | 0 | 0
Period: 1st Cycle of Maintenance (3 Weeks)
Arm/Group | Brentuximab Vedotin Dose Level -1 (0.8 mg/kg) | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Started | 0 | 20 (Consolidation is optional for patients who have a partial or complete response during induction)
Received Dose of Study Drug | 0 | 14
Completed | 0 | 14
Not Completed | 0 | 6
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1
Period: 2nd Cycle of Maintenance and Beyond
Arm/Group | Brentuximab Vedotin Dose Level -1 (0.8 mg/kg) | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Started | 0 | 14
Received Dose of Study Drug | 0 | 14
Completed (Completion = up to 1 year of maint. treatment from time of induction (1 maint. cycle = 3 weeks).) | 0 | 2
Not Completed | 0 | 12
Not completed — Adverse Event | 0 | 10
Not completed — Progressive Disease | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Follow Up (up to 3 Years)
Arm/Group | Brentuximab Vedotin Dose Level -1 (0.8 mg/kg) | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Started | 0 | 20 (Patients who received at least one dose of study treatment go into follow-up.)
Completed | 0 | 14
Not Completed | 0 | 6
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: For Phase I: The Recommended Phase 2 Dose of Brentuximab Vedotin in Combination With Rituximab.
Description: To identify the recommended phase 2 dose (RP2D)/maximum tolerated dose (MTD) of brentuximab vedotin in combination with rituximab. The dose limiting toxicity monitoring period for brentuximab vedotin and rituximab is first 21 days (during induction).The RP2D/MTD will be defined as the highest dose of brentuximab vedotin that causes dose limiting toxicities (DLTs) in <2 of 6 patients. The Phase I portion of the study follows a 3+3 design. Brentuximab has two dose levels: Level 1 (starting dose) 1.2 mg/kg IV, and Level -1 (de-escalation dose): 0.8 mg/kg IV. Toxicity will be assessed using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 4.03.
Time Frame: The first 21 days of Induction
Measure: Number; unit: mg/kg
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 6
mg/kg | 1.2

2. Primary Outcome: Phase 1: Number of Dose Limiting Toxicities of Brentuximab Vedotin and Rituximab in Patients With Immunosuppressed Lymphoid Malignancies.
Description: Dose limiting toxicities (DLT) will be monitored for Phase 1 patients for the first 21 days of Induction (the DLT monitoring period) to evaluate safety. In general, a non-hematologic DLT is defined as any Grade ≥ 3 toxicity, and a hematologic DLT is defined as any Grade ≥ 4 toxicity, both by CTCAE v4.03 criteria.
Time Frame: The first 21 days of induction
Population: Six patients in Phase 1 received dose level 1 of brentuximab vedotin (1.2 mg/kg IV).
Measure: Number; unit: Grade 3 hyponatremia
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 6
Grade 3 hyponatremia | 1

3. Primary Outcome: Phase II: Percent of Participants With an Overall Response
Description: Overall response will be defined as the detection of Partial Response (PR) or Complete Response (CR) by CT or PET/CT, and/or resolution of marrow-only involvement. Response will be assessed according to the Revised Response Criteria for Malignant Lymphoma (Cheson, et al). CR is defined as a complete disappearance of all detectable clinical evidence of disease and disease-related symptoms, if present before therapy. A post-treatment residual mass of any size is permitted as long as it is PET negative. If a pretreatment PET scan was negative, all lymph nodes and nodal masses must have regressed on CT to normal size. A PR is defined as At least a 50% decrease in sum of the product of the diameters of up to six of the largest dominant nodes or nodal masses. No increase should be observed in the size of other nodes, liver, or spleen.
Time Frame: Every 12 weeks for up to 1 year on treatment (Range of cycles attempted from induction, +/- consolidation, + maintenance = 1-17 cycles) Induction = 4 weeks, consolidation = 4 weeks, 1 maintenance cycle = 3 weeks
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 20
percent of participants | 75 [51 to 91]

4. Secondary Outcome: Number of Participants With Adverse Events Possibly Related to Study Drug Graded 3, 4, and 5
Description: Toxicity, both frequency and severity, will continue to be measured by monitoring the occurrence of adverse events. Adverse events will be defined as those included in CTCAE v 4.03. AEs that were determined to be at least possibly related to study drug and graded 3, 4, 5 are included here. Grade 1 (mild): the event causes discomfort without disruption of normal daily activities. Grade 2 (moderate): the event causes discomfort that affects normal daily activities. Grade 3 (severe): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status. Grade 4 (Life-threatening): the patient was at risk of death at the time of the event. Grade 5 (fatal): the event caused death.
Time Frame: From time of treatment to 30 days post discontinuation (range of cycles attempted from induction +/- consolidation, & maintenance = 1-17 cycles) About 1 year Induction = 4 weeks, consolidation = 4 weeks, 1 maintenance cycle = 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 20
Participants
  Grade 3 Diarrhea | 1
  Grade 4 Hyperbilirubinemia | 1
  Grade 3 AST elevation | 2
  Grade 4 Lipase elevation | 2
  Grade 3 Amylase elevation | 1
  Grade 4 Amylase elevation | 1
  Grade 4 Typhlitis | 1
  Grade 3 Anemia | 2
  Grade 3 Febrile Neutropenia | 1
  Grade 3 Lymphopenia | 7
  Grade 4 Lymphopenia | 2
  Grade 4 Neutropenia | 1
  Grade 3 Neutropenia | 7
  Grade 3 Elevated creatinine | 1
  Grade 3 Acute kidney injury | 2
  Grade 3 Hypophosphatemia | 1
  Grade 3 Peripheral neuropathy | 2

5. Secondary Outcome: Percentage of Participants Without Progression (Progression Free Survival (PFS))
Description: Study treatment efficacy will be evaluated using PET or CT scan images to determine Progression Free Survival (PFS). PFS is defined as the duration of time from start of treatment to time of progression. Response criteria will be those specified by Cheson, et al as the Revised Response Criteria for Malignant Lymphoma. Progressive Disease (PD) is defined as the appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size, or at least a 50% increase from nadir in the diameter of any previously involved nodes, or in a single involved node, or the size of other lesions. All patients who have had at least one dose of study treatment will be evaluable for PFS with censoring of patients who are lost to follow-up. PFS will be reported as percentage of participants without progression.
Time Frame: start of treatment to time of progression (up to 2 years after treatment discontinuation)
Population: One patient was excluded from the analysis because they were lost to follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 19
percentage of participants | 75 [52 to 96]

6. Secondary Outcome: Percentage of Participants Alive at 2 Years (Overall Survival)
Description: Overall survival (OS) will be measured from treatment initiation until death from any cause for up to 1 year post-treatment discontinuation. Overall survival is defined as the duration of time from start of treatment to time of death. All patients who have had at least one dose of study treatment will be evaluable for OS. OS will be reported as percentage of participants alive at 2 years post treatment discontinuation, with censoring of patients who are lost to follow-up.
Time Frame: From start of treatment to 2 years post treatment discontinuation
Population: One patient was censored from overall survival because they were lost to follow-up.
Measure: Number (90% Confidence Interval); unit: percent of participants
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 19
percent of participants | 90 [77 to 100]

7. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: The best overall response (BOR) is the best response recorded from the start of the treatment until disease progression/recurrence. Best response assessed by CT or PET/CT according to the Revised Response Criteria for Malignant Lymphoma (Cheson et. al). Responses include Complete Response (CR), Partial Response (PR), and Stable Disease (SD). CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms, if present before therapy. If a pretreatment PET scan was negative, all lymph nodes and nodal masses must have regressed on CT to normal size. PR: At least a 50% decrease in sum of the product of the diameters of up to six of the largest dominant nodes or nodal masses. No increase should be observed in the size of other nodes, liver, or spleen. SD: neither CR or PR, or progressive disease (PD). PD: Appearance of new lesion > 1.5 cm in any axis, or at least a 50% increase from nadir in the diameter of any previously involved nodes.
Time Frame: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 20
participants
  Complete Response | 12
  Partial Response | 3
  Stable Disease | 3

8. Secondary Outcome: Number of Participants With Epstein Barr Virus (EBV) Activation and Number of Participants Without EBV Activation
Description: EBV activation will be evaluated in all patients who receive at least one dose of study treatment and have an evaluable tissue microarray (TMA) collected at baseline. EBV activation and proliferation will be measured by viral loads from blood collections as measured at time of enrollment and monthly thereafter in all enrolled patients, until completion of study therapy. Epstein Barr Virus (EBV) quantitative PCR is used to an aid in monitoring EBV-related disease. Lab thresholds vary at sites however, labs results are considered either "negative" or "abnormal". Number of participants who experienced EBV activation, i.e an abnormal lab result (YES) and patients who did not experience EBV activation, i.e. a negative lab result (NO) will be reported.
Time Frame: Time from start of study treatment to last dose of study drug (Range of cycles attempted from induction, +/- consolidation, + maintenance = 1-17 cycles, up to 1 year) Induction = 4 weeks, consolidation = 4 weeks, 1 maintenance cycle = 3 weeks
Population: 1 patient was not evaluable. They withdrew consent before data could be collected.
Measure: Number; unit: participants
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 19
participants
  EBV Activation: YES | 1
  EBV Activation: NO | 18

9. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy
Description: Time to initiation of cytotoxic chemotherapy will be defined as the time elapsed between study treatment initiation, and time of first non-targeted cytotoxic chemotherapy (off study treatment). Time to cytotoxic chemotherapy will be evaluated in all patients who receive at least one dose of study treatment.
Time Frame: Up to 3 years from treatment discontinuation
Population: Follow-up data for time to initiation of cytotoxic chemotherapy was collected for only 5 patients. That data is reported below.
Measure: Number; unit: number of days
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 5
number of days
  Patient 1 | 35
  Patient 2 | 147
  Patient 3 | 38
  Patient 4 | 184
  Patient 5 | 66

10. Secondary Outcome: Number of Participants With Graft Rejection vs Without Graft Rejection
Description: Graft rejection will be defined as any of the following: documentation of new or progressive rejection by tissue biopsy of the graft; re-transplantation due to graft rejection; clinical diagnosis of new or progressive graft rejection, since start of treatment on protocol, as given by the patient's transplant physician. Escalation of intensity of immunosuppression will not, by itself, be considered evidence of graft rejection. Note: patients with clinically active graft rejection will not be excluded from trial enrollment, but will not be considered to have treatment emergent graft rejection unless progression of rejection is documented. Rates of graft rejection will be evaluated in all patients who receive at least one dose of study treatment.
Time Frame: From start of treatment to 3 years post treatment discontinuation
Population: 1 patient was not evaluable. They withdrew consent before data could be collected.
Measure: Number; unit: participants
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 19
participants
  Graft Rejection: YES | 1
  Graft Rejection: NO | 18

11. Post Hoc Outcome: Median Time to Best Response
Description: Time to best response = the number of days from treatment initiation to best response (complete response/CR or partial response/PR). Best response assessed by CT or PET/CT according to the Revised Response Criteria for Malignant Lymphoma (Cheson et. al). Responses include Complete Response (CR), Partial Response (PR), and Stable Disease (SD). CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms, if present before therapy. If a pretreatment PET scan was negative, all lymph nodes and nodal masses must have regressed on CT to normal size. PR: At least a 50% decrease in sum of the product of the diameters of up to six of the largest dominant nodes or nodal masses. No increase should be observed in the size of other nodes, liver, or spleen. SD: neither CR or PR, or progressive disease (PD). PD: Appearance of new lesion > 1.5 cm in any axis, or at least a 50% increase from nadir in the diameter of any previously involved nodes.
Time Frame: From start of treatment, every 12 weeks for up to 1 year on treatment (Range of cycles attempted from induction, +/- consolidation, + maintenance = 1-17 cycles) Induction = 4 weeks, consolidation = 4 weeks, 1 maintenance cycle = 3 weeks
Measure: Median (Full Range); unit: number of days
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
Number analyzed (Participants) | 20
number of days | 28 [23 to 151]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 5 year period. Each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 30 days post last treatment. Induction = 28 days, consolidation (optional) = 28 days, 1 maintenance cycle = 21 days, with treatment lasting up to 1 year from induction. The range of cycles attempted was 1-17 (including induction +/- consolidation, and maintenance).
Description: Brentuximab vedotin dose level -1 (dose de-escalation level) never opened. All 20 patients received dose level 1 (1.2 mg/kg) of brentuximab vedotin.
Arm/Group | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg)
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 14/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg) (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lung Infection (Infections and infestations) | 2 — 1 patient also experienced dyspena and chest pain at the time of this event. 1 patient also experienced upper respiratory infection at the time of this event.
Neutrophil count decreased (Investigations) | 1 — 1 patient also experienced fever at the time of this event.
Acute kidney injury (Renal and urinary disorders) | 2 — 1 patient also experienced chills and malaise at the time of this event.
Abdominal pain (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 1
Sepsis (Infections and infestations) | 2 — 1 patient also experienced a decrease in neutrophil count at the time of this event.
Dehydration (Metabolism and nutrition disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Fatigue (General disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 1 — This patient also experienced hyperglycemia, pneumonia, drug-induced liver injury, and catheter-associated urinary tract infection at the time of this event.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximb Vedotin Dose Level 1 (1.2 mg/kg) (N=20)
Anemia (Blood and lymphatic system disorders) | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Heart murmur (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 4
Ventricular arrhythmia (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 1
Cataract (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Floaters (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Enterocolitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Abnormal satiety (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Oral pain (Gastrointestinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Chills (General disorders) | 2
Edema face (General disorders) | 1
Edema limbs (General disorders) | 7
Fatigue (General disorders) | 10
Fever (General disorders) | 6
Night sweats (General disorders) | 2
Infusion related reaction (General disorders) | 2
Injection site reaction (General disorders) | 1
Irritability (General disorders) | 1
Malaise (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 7
Cholecystitis (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Systemic inflammatory response syndrome (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Swollen ankle (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 5
Creatinine increased (Investigations) | 11
INR increased (Investigations) | 3
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 18
Neutrophil count decreased (Investigations) | 10
Platelet count decreased (Investigations) | 8
Serum amylase increased (Investigations) | 4
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 10
Acidosis (Metabolism and nutrition disorders) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hyperkalemia (Metabolism and nutrition disorders) | 8
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Sessile polyp in descending colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 5
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Memory impairment (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Altered mental state (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 7
Hematuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Elevated liver enzymes (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Benign paroxysmal positional vertigo (Nervous system disorders) | 1
Difficulty with fine motor skills (Nervous system disorders) | 1
Restless leg syndrome (Nervous system disorders) | 1
Increase urinary frequency (Renal and urinary disorders) | 2
Malodorous urine (Renal and urinary disorders) | 1
Low glomerular filtration rate (Renal and urinary disorders) | 1
Renal tubulitis (Renal and urinary disorders) | 1
Catheter associated urinary tract infection (Renal and urinary disorders) | 1
Polyp underneath eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Platelet count increased (Investigations) | 1
Abnormal Blood Urea Nitrogen (Investigations) | 2
Increased Lactate Dehydrogenase (Investigations) | 1
Decreased monocytes (Investigations) | 1
Generalized body soreness (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Muscle twinges in legs, abdomen, and chest (Musculoskeletal and connective tissue disorders) | 1
Left shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Hypovolemia (Metabolism and nutrition disorders) | 1
Low iron (Metabolism and nutrition disorders) | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 1
Mouth sores (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Worsening of right lung opacity in CT scan (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Shortness of breath with exertion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Itching of medial portion of the knees (Skin and subcutaneous tissue disorders) | 1
tender back (Skin and subcutaneous tissue disorders) | 1
redness of left leg (Skin and subcutaneous tissue disorders) | 1
Cellulitis behind ear (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study did not meet it's accrual goal of 33 patients. The study closed due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT01805037/Prot_SAP_000.pdf